CLINICAL TRIAL: NCT03444389
Title: An Investigation Into the Relationship Between Hemorrhoid Disease and the Use of Smartphones in the Lavatory
Brief Title: The Relationship Between Hemorrhoids and Smartphone Use in the Lavatory
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Sebahattin Celik, Assistant Professor, Department of General Surgery, Yuzuncu Yil University
Other Study IDs: 12/22/2017- 051
Record Dates: First submitted 2018-01-31; First posted 2018-02-23 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Patients with hemorrhoids
- Control group: Healthy participants without hemorrhoids

SUMMARY:
The objective of this study is to examine the relationship between hemorrhoids, a common complaint, and the use of smartphones, also a common feature of modern life, in the lavatory.

As is known, hemorrhoidal disease is a frequently observed disease of the lower rectum and anal region that seriously impairs the patient's quality of life.

Based on clinical observations, the study investigators have found that the use of mobile phones in the lavatory has become a habit for some people. The investigators surmise that this habit, which increases the time spent on the toilet, also leads to an increase in pressure on the anal region and straining during defecation. There is a gap in the literature investigating the relationship between these two situations (smartphone use in the lavatory and the development of hemorrhoids). The basic research question of the present study is thus designed to determine to what extent the use of smartphones increases time spent in the lavatory and whether there is an association between this increase in time and hemorrhoidal disease.

DETAILED DESCRIPTION:
The objective of this study is to examine the relationship between hemorrhoids, a common complaint, and the use of smartphones, also a common feature of modern life, in the lavatory.

As is known, hemorrhoidal disease is a frequently observed disease of the lower rectum and anal region that seriously impairs the patient's quality of life. The underlying pathophysiological event is vascular enlargement of the lower rectum. Hemorrhoids are classified as internal or external, and it is assumed that the same pathological mechanisms operate in both types. Accepted pathological mechanisms and predisposing factors of hemorrhoids include reduced venous drainage, straining while defecating, constipation, pregnancy, portal hypertension and anorectal varices, and other risk factors.

Given the pathophysiological and accelerating factors described above, an increase in hemorrhoidal disease in modern society is to be expected. People today prefer a more sedentary lifestyle and partake of a low-fiber diet richer in high calorie/high fat foods compared with previous generations. In addition, smartphones have invaded nearly every aspect of daily life. Based on clinical observations, the investigators have found that the use of mobile phones in the lavatory has become a habit for some people. The investigators surmise that this habit, which increases the time spent on the toilet, also leads to an increase in pressure on the anal region and straining during defecation. There is a gap in the literature investigating the relationship between these two situations (smartphone use in the lavatory and the development of hemorrhoids), and researching this relationship could reveal important information. The basic research question of the present study is thus designed to determine to what extent the use of smartphones increases time spent in the lavatory and whether there is an association between this increase in time and hemorrhoidal disease.

This clinical study will be conducted with a cross-sectional design based on retrospective observation. Apart from the target population there will be a control group. In retrospective studies the selection of the control group is of the utmost importance. Other than the risk factor that is being investigated (the use of smartphones), factors that affect the development of hemorrhoid disease are similar for the study group and the control group, thus minimizing confounding factors. The control group, as will be noted, will thus have a social environment resembling that of the study group. It should also be noted that members of the control group will be completely healthy, with no health problems (e.g., hearing or visual disturbances) that could affect their use of the risk factor (smartphones).

The study population consists of patients with complaints of hemorrhoids referred to the General Surgery Polyclinic. The control group is comprised of healthy volunteers with no complaints of hemorrhoids. Both the study group and the control group will include persons of both genders between 16 and 65 years of age. Informed consent will be obtained from patients and volunteers, following which a Likert-type survey will be given to each participant to complete. A pilot study will be conducted for the factor analysis of the questions to be asked in the questionnaire. In the pilot study, the target will be to survey 100 patients. After the factor analysis is performed on 100 patients, the questionnaire that is developed will be used in the main study.

As no prevalence study was previously performed for the sample size, it will be calculated based on the prevalence (frequency of smartphone use in the lavatory in the study group and the control group) determined after the pilot study, by accepting a type I error of 0.05 and a type II error of 0.20 (80% test power).

The doctor who performs the examinations will be blinded to the questionnaire results. After completion of the questionnaire, the patient's anal region and rectum will be examined by a general surgeon and the presence or absence of hemorrhoids will be noted. Subsequently, if hemorrhoids are present, they will be recorded as either external or internal. Internal hemorrhoids will then be staged as first-degree, second-degree, third-degree, or fourth-degree, according to the standard textbook definitions.

ELIGIBILITY:
Inclusion Criteria:

* The study group consists of people with hemorrhoids.
* The control group consists of healthy participants without hemorrhoids.
* The study and control groups should have similar habits in terms of lifestyle, eating habits, etc.

Exclusion Criteria:

* The control group participants should have no vision, hearing, or other problems that restrict or otherwise affect their use of smartphones (the risk factor).
* Participants should not have health problems that may be a causative factor in the pathogenesis of hemorrhoids.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with complaints of hemorrhoids who were referred to the General Surgery Polyclinic.
Sampling Method: Non-Probability Sample
Enrollment: 1798 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of hemorrhoids | Through study completion (up to 7 months)
  A physical examination is performed by a general surgeon to determine presence or absence of hemorrhoids.

SECONDARY OUTCOMES:
Degree of hemorrhoids (if present) | Through study completion (up to 7 months)
  A physical examination is performed by a general surgeon to determine degree (1st to 4th) of hemorrhoids.
Smartphone usage habits in the lavatory | Through study completion (up to 7 months)
  A questionnaire is used to investigate the relationship between smartphone use in the lavatory and hemorrhoid disease. The desired measure is the total amount of time (in minutes) that smartphone use in the lavatory increases time spent in the lavatory each day. This measure is based on the answers to two questions: the number of times per day that the participant uses the lavatory for defecation (1; 2; 3; 4; 5-10; more than 10), multiplied by the length of time that lavatory visits are increased due to smartphone use (no choices are given; instead, the participant enters the number of minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Sebahattin Celik, M.D., Principal Investigator — Department of General Surgery, Yuzuncu Yil University Faculty of Medicine
Locations (1):
- Yuzuncu Yil University Faculty of Medicine, Van, Turkey (Türkiye)

REFERENCES:
- [Background] Haas PA, Haas GP, Schmaltz S, Fox TA Jr. The prevalence of hemorrhoids. Dis Colon Rectum. 1983 Jul;26(7):435-9. doi: 10.1007/BF02556521. PMID 6861574
- [Background] Fox A, Tietze PH, Ramakrishnan K. Anorectal conditions: hemorrhoids. FP Essent. 2014 Apr;419:11-9. PMID 24742083
- [Background] Gibbons CP, Bannister JJ, Read NW. Role of constipation and anal hypertonia in the pathogenesis of haemorrhoids. Br J Surg. 1988 Jul;75(7):656-60. doi: 10.1002/bjs.1800750712. PMID 3416121
- [Background] Johanson JF, Sonnenberg A. The prevalence of hemorrhoids and chronic constipation. An epidemiologic study. Gastroenterology. 1990 Feb;98(2):380-6. doi: 10.1016/0016-5085(90)90828-o. PMID 2295392
- [Background] Johanson JF, Sonnenberg A. Constipation is not a risk factor for hemorrhoids: a case-control study of potential etiological agents. Am J Gastroenterol. 1994 Nov;89(11):1981-6. PMID 7942722
- [Background] Wald A. Constipation, diarrhea, and symptomatic hemorrhoids during pregnancy. Gastroenterol Clin North Am. 2003 Mar;32(1):309-22, vii. doi: 10.1016/s0889-8553(02)00069-9. PMID 12635420
- [Background] Staroselsky A, Nava-Ocampo AA, Vohra S, Koren G. Hemorrhoids in pregnancy. Can Fam Physician. 2008 Feb;54(2):189-90. PMID 18272631
- [Background] Gojnic M, Dugalic V, Papic M, Vidakovic S, Milicevic S, Pervulov M. The significance of detailed examination of hemorrhoids during pregnancy. Clin Exp Obstet Gynecol. 2005;32(3):183-4. PMID 16433160
- [Background] Bernstein WC. What are hemorrhoids and what is their relationship to the portal venous system? Dis Colon Rectum. 1983 Dec;26(12):829-34. doi: 10.1007/BF02554764. PMID 6605842
- [Background] Misra SP, Dwivedi M, Misra V. Prevalence and factors influencing hemorrhoids, anorectal varices, and colopathy in patients with portal hypertension. Endoscopy. 1996 May;28(4):340-5. doi: 10.1055/s-2007-1005477. PMID 8813499
- [Background] Lowney JK, Fleshman JW Jr. Benign disorders of the anorectum (pelvic floor, fissures, hemorrhoids, and fistulas). In: Zinner MJ, Ashley SW, eds. Maingot's Abdominal Operations. 11th ed. New York: McGraw-Hill; 2007: 663-693.

DOCUMENTS (3):
  • Study Protocol (2018-02-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03444389/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT03444389/SAP_001.pdf
  • Informed Consent Form (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT03444389/ICF_002.pdf